CLINICAL TRIAL: NCT03988127
Title: Validation of Perfusion Index as a Tool for Pain Assessment in Critically Ill Intubated Patients
Brief Title: Perfusion Index in Pain Assessment
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Kamal Zahran, Principal Investigator, Cairo University
Other Study IDs: S-8-2019
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Perfusion index — The perfusion index (PI) is the ratio of the pulsatile to the non-pulsatile blood flow in peripheral tissue. It represents a non-invasive measure of peripheral perfusion that can be continuously obtained from a pulse oximeter. We observe changes in PI before and after painful stimulation in intubated critically ill patients.

SUMMARY:
The perfusion index (PI) is the ratio of the pulsatile to the non-pulsatile blood flow in peripheral tissue. It represents a non-invasive measure of peripheral perfusion that can be continuously obtained from a pulse oximeter. This property explains the fact that it decreases with vasoconstriction and increases with vasodilatation.

An increase in PI was proved to be an early indicator for the success of general and regional anaesthesia, which cause initial peripheral vasodilatation before the onset of anaesthetic effect. Whereas a failed increase in PI would suggest failure of anaesthesia.

The PI has been reported to decrease when noxious stimulus was applied to anaesthetized volunteers. A recent study on critically ill non-intubated patients has demonstrated a good correlation between changes in PI and changes in Behavioral Pain Scale-non intubated values after a painful stimulus was applied.

Despite the rising use of perfusion index in anaesthesia and intensive care, few studies have investigated its capability as a pain assessment tool, and to our knowledge, it has not been investigated in intubated critically ill patients yet.

DETAILED DESCRIPTION:
All patients after admission will be monitored with the use of routine monitoring tools: Electrocardiogram, pulse oximetry, and automated noninvasive blood pressure (NIBP). Day-to-day investigations will be carried out to monitor and individualize treatment. Medical (and/or) surgical treatment will be performed, supervised by the attending intensivist and surgeon.

Sedation and analgesia protocol will be prescribed by the patient's primary intensivist. Another pulse oximeter probe (Masimo Radical 7; Masimo Corp., Irvine, CA, USA) will be attached to the patient's index finger during changing the patient's position (head of bed elevation) after abdominal surgery. This pulse oximeter will be connected to the Masimo monitor and shielded to prevent outside light from interfering with the signal.

Sedation will be assessed by using the Richmond Agitation- Sedation scale (RASS). Pain assessment will be achieved by using the behavioural pain scale intubated (BPS-IN).

Sedation and analgesia will be guided by the BPS and RASS. For analgesia the patients will receive a loading dose (0.05-0.2 mg/kg) morphine sulphate I.V., followed by (2-10 mg/h) infusion to keep the BPS between 3 and 6. If the pain score is more than 6, a rescue dose of 3 mg will be given, and then the pain will be reassessed after 5 min. If the patient received more than 2 boluses/h, the infusion dose will be increased by 2 mg/h.

For sedation, the patients will receive a loading dose of propofol 0.005 mg/kg/min IV for at least 5 min., followed by (0.005-0.05 mg/kg/min) IV infusion to achieve a RASS score of 0 to -1. A rescue dose of 5-10 mcg/kg/min over 5-10 min intervals if the RASS score is more than 0; allow a minimum of 5 min between adjustments for onset of peak effect.

ELIGIBILITY:
Inclusion Criteria:

* Sedated intubated surgical ICU patients during the first two postoperative days following abdominal surgery.

Exclusion Criteria:

* Patients with a history of neurologic disorder (hemiparesis, quadriparesis, and neuropathy).
* Patients with an epidural catheter with local anaesthetic injection for the purpose of analgesia.
* Patients receiving neuromuscular blockade.
* Patients with peripheral vascular disease.
* Patients suffering from fever.
* Hypothermia.
* Use of vasopressors.
* Patients with altered level of consciousness (GCS <4).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sedated intubated surgical ICU patients aged 18 to 60 years old
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
The correlation between delta PI and delta BPS | 1 minute before the painful stimulus and 1 minute after.
  We observe the correlation between the changes in Perfusion index vales and the changes in Behavioral Pain Scale vales before and after the application of painful stimulus

SECONDARY OUTCOMES:
Systolic blood pressure | 1 minute before the painful stimulus and 1 minute after.
  mmHg
Diastolic blood pressure | 1 minute before the painful stimulus and 1 minute after.
  mmHg
Heart rate | 1 minute before the painful stimulus and 1 minute after.
  beat per minute
Richmond Agitation- Sedation scale | 1 minute before the painful stimulus and 1 minute after.
  * 4: Combative
  * 3: Very agitated
  * 2: Agitated
  * 1: Restless 0: Alert and calm
    * 1: Drowsy
    * 2: Light sedation
    * 3: Moderate sedation
    * 4: Deep sedation
    * 5: Unarousable
Sensitivity and specificity of PI to predict BPS > or = 6 | 1 minute before the painful stimulus and 1 minute after.
  By generating Receiver Operating Characteristic curve

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided